CLINICAL TRIAL: NCT00299026
Title: TAXUS II: A Randomized, Double-Blind, Controlled Study of the Safety and Performance of the NIRx™ Paclitaxel-Coated Conformer Coronary Stent
Brief Title: A Randomized, Double-Blind, Controlled Study of the Safety and Performance of the NIRx™ Paclitaxel-Coated Conformer Coronary Stent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Thomas Naeschen, PhD, Boston Scientific
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAXUS II; S2003
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Stent Implant; Drug-coated Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NIRx(TM) Paclitaxel-Coated Conformer Coronary Stent System

SUMMARY:
The clinical investigation is an international, prospective, double-blind, randomized safety and efficacy study. The purpose of this study is to evaluate the safety and performance of the NIRx(TM) Paclitaxel-Coated Stent (1.0µg/mm2 of paclitaxel incorporated into slow- and moderate-release formulation of a triblock copolymer carrier system)in patients who present for stenting of de novo lesions of a native coronary artery.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and performance of coronary artery stenting with the NIRx(TM) Paclitaxel-Coated Stent (1.0µg/mm2 of paclitaxel incorporated into slow- and moderate-release formulation of a triblock copolymer carrier system) for the treatment of de novo lesions in native vessels. Patients in 2 sequential cohorts will be randomised to receive either the NIRx(TM) Paclitaxel-Coated Stent or the uncoated control stent. In cohort 1, the slow-release formulation NIRx(TM) Paclitaxel-Coated Stent will be studied. If the safety profile is acceptable, the moderate-release formulation NIRx(TM) Paclitaxel-Coated Stent will be studied in Cohort 2. In each f the 2 cohorts, 133 patients will be treated with the NIRx(TM) paclitaxel-Coated Stent and 133 with the uncoated control stent (1.1 ratio), for a total of 532 patients in study.

ELIGIBILITY:
General Inclusion Criteria:

* Patient >= 18 years old.
* Eligible for percutaneous transluminal coronary angioplasty (PTCA).
* Patient (or legal guardian) understands the study requirements and the stent treatment procedure and provides written Informed Consent before any study-specific tests or procedures are performed.
* Willing to comply with all specified follow-up evaluations.
* Documented stable angina pectoris (Canadian Cardiovascular Society Classification [CCS] 1, 2, 3, or 4), unstable angina pectoris with documented ischemia (Braunwald Class IB - C, IIB - C, or IIIB - C), or documented silent ischemia.
* Acceptable candidate for CABG.

Angiographic Inclusion Criteria:

* Target lesion is located within a native coronary vessel.
* Target lesion is de novo (i.e., a coronary lesion not previously treated).
* Target lesion diameter stenosis >= 50% and <= 99% (visual estimate or on-line QCA).
* Target lesion <= 12 mm in length (visual estimate or on-line QCA).
* Target vessel >= 3.0 mm and <= 3.5 mm in diameter (visual estimate or on-line QCA).

General Exclusion Criteria:

* Known sensitivity to paclitaxel.
* Patient has received paclitaxel or other anti-mitogenic agent within 12 months prior to planned enrollment in the study.
* Patient has previous stent procedure with any drug-coated or drug-eluting stent device.
* Patient has undergone any coronary intervention within 30 days prior to stent placement associated with this protocol.
* Patient anticipates planned additional intervention (staged procedure) to any non-target coronary vessel within 45 days after the stent placement associated with this protocol.
* MI within 72 hours of planned stent placement.
* Left ventricular ejection fraction (LVEF) of < 30%.
* Stroke within the past 6 months.
* Acute or chronic renal dysfunction (creatinine >1.7 mg/mL or >150 µmol/L).
* Acetylsalicylic acid and/or clopidogrel and/or ticlopidine are contraindicated.
* Leukopenia (leukocytes <3.5 x 109/liter).
* Thrombocytopenia (platelets <100,000/mm3).
* Active peptic ulcer or active gastrointestinal (GI) bleeding.
* Known allergy to stainless steel.
* Previously enrolled in the NIRx(TM) Coronary Stent Clinical Safety and Performance Study.
* Currently enrolled in another investigational device or drug study and has not completed the required follow-up period, or has completed all other study-required follow-up less than 30 days prior to enrollment in this study.
* Patient is lactating, has a positive pregnancy test within 7 days of planned stent placement, or intends to become pregnant during the study (only applies to female patients of child-bearing potential).
* Life expectancy of less than 24 months because of other medical conditions.
* Co-morbid condition(s) that could limit the patient's ability to participate in the study or comply with follow-up requirements or co-morbid condition(s) that could impact the scientific integrity of the study.

Angiographic Exclusion Criteria:

* Unprotected left main coronary artery disease (or obstruction greater than 50% in the left main coronary artery that is not protected by at least 1 non-obstructed bypass graft to the left anterior descending [LAD] or circumflex artery or a branch thereof).
* Target lesion is in a previously stented segment.
* Target vessel was treated with directional coronary atherectomy, laser, or transluminal extraction catheter prior to stent placement.
* Target lesion is ostial in location (within 3 mm of vessel origin).
* Target site of stent placement has side branches >2.0 mm in diameter.
* Target lesion is severely calcified (by visual estimate)
* Target vessel has closed abruptly or is threatening closure.
* Target lesion is located within or immediately distal to a >60° bend in the vessel.
* Target vessel has diffuse disease requiring more than one 15 mm stent for full lesion coverage.
* Target lesion involves a bifurcation where a branch vessel greater than 2.0 mm in diameter originates (either stenosis of both main vessel and major branch or stenosis of just major branch).
* Target lesion has excessive tortuosity unsuitable for stent delivery and deployment.
* Target lesion is located within a saphenous vein bypass graft.
* Target lesion is located in a vessel section supplied by distal graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532
Dates: Start 2001-06; Primary Completion 2003-05 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Mean percent in-stent net volume obstruction at 6 months post-procedure as measured by IVUS

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — Ospedale San Raffaele del Monte Tabor
Locations (1):
- San Raffaele del Monte Tabor, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silber S, Colombo A, Banning AP, Hauptmann K, Drzewiecki J, Grube E, Dudek D, Baim DS. Final 5-year results of the TAXUS II trial: a randomized study to assess the effectiveness of slow- and moderate-release polymer-based paclitaxel-eluting stents for de novo coronary artery lesions. Circulation. 2009 Oct 13;120(15):1498-504. doi: 10.1161/CIRCULATIONAHA.109.849877. Epub 2009 Sep 28. PMID 19786634